CLINICAL TRIAL: NCT06607484
Title: Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Effects of SR-878 in Healthy Volunteers
Brief Title: Study Investigating the Safety, Tolerability and Blood Concentration of the Substance SR-878
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: SciRhom GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SR-878-01-001; 2023-507753-15-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-04; First posted 2024-09-23 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SR-878 (Experimental): Solution for infusion, administered intravenously once
  Interventions: Drug: SR-878
- Placebo (Placebo Comparator): Solution for infusion, administered intravenously once
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SR-878 — Intravenous infusion
  Arms: SR-878
Drug: Placebo — Intravenous infusion
  Arms: Placebo

SUMMARY:
SR-878 is a newly developed medicine that aims to treat autoimmune disorders. It inhibits a protein (iRhom2), that regulates enzymes that are involved in the production of cytokines (small proteins that are crucial in controlling the activity of immune system cells). This is the first study in humans, and SR-878 will be administered once to each participant in 6 different doses to establish a safe dosage and investigate, what are potential side effects.

This clinical trial includes six study groups, called cohorts, and each cohort includes 8 participants. In each cohort, 6 participants will receive SR-878 and 2 participants will receive a placebo, a dummy drug with no active ingredients that looks identical. The comparison with placebo will be used to better assess the side effects of SR-878. The dose of SR-878 will be gradually increased between cohorts. Participants in the first cohort will receive the lowest dose, and if this is considered safe 10 days after dosing, the next cohort will be initiated at a higher dose. Participants visit the hospital regularly over the next 12 weeks after receiving SR-878 or placebo. During these visits, medical condition will be checked and blood will be taken.

Participants in the third to sixth cohort will be injected with a product called LPS 24 hours after the infusion of the investigational product, which may stimulate the immune system and cause a temporary inflammatory response in the body. During this time, participants may have mild "flu-like" symptoms. 12 weeks after dose of investigational product, the LPS injection and saline infusion will be repeated.

DETAILED DESCRIPTION:
Rationale: SR-878 is a newly developed medicine that aims to treat autoimmune disorders. It works by blocking a protein called iRhom2, which controls the production of small proteins called cytokines. Cytokines are the drivers that keep the inflammatory process ongoing in autoimmune diseases important for regulating the activity of cells in the immune system. This is the first study in humans, and SR-878 will be administered once to each participant in 6 different doses to investigate potential side effects.

Objectives:

* To assess the safety and tolerability of a single dose of SR-878;
* To select the optimal dose that is safe and tolerable;
* To explore any effects of a single dose of SR-878 in the human body;
* To investigate the connection between the concentration of SR-878 and potential side effects;
* To assess the amount of immune response against SR-878. Trial design: This clinical study will have six treatment groups, so called cohorts, and each cohort will include 8 participants. In each cohort 6 participants will receive SR-878, and 2 participants will receive a placebo, that is a dummy treatment without active ingredients. The comparison with the placebo is used to better assess the side effects of SR-878. The dose of SR-878 will be gradually increased between cohorts.

After the screening period, participants will be randomly assigned to receive SR-878 or placebo. This is a double-blind study, which means neither the participant nor the study staff, including the study doctor, will know which study medication was used.

The study medication will be administered in a 1-hour long infusion. The participants will be requested to stay 24 hours in the hospital after the infusion, and their medical condition will be monitored, and they will undergo several blood draws.

24 hours after the study medication infusion, participants in the 3rd-6th cohorts, will be injected with a product, called lipopolysaccharide (LPS). It has the ability to boost the body's immune response, even without causing an actual infection. LPS might trigger slight flu-like symptoms (i.e. uneasiness, little fever). Participants will be requested to stay an additional 8 hours in the hospital, and they will undergo several blood samplings and their body's reaction will be monitored. In the first 6 hours, they will receive a saline infusion to keep them hydrated, and in case they find the potential symptoms of the provoked inflammation unbearable, the study doctor will provide a medication (paracetamol) to relieve them.

In the following 12 weeks, participants will be requested to return regularly to the hospital, 10 times in total. During these visits, their medical status will be examined, and blood will be collected. For participants in the 3rd-6th cohorts, 12 weeks after their study medication dose, the LPS injection and the saline infusion will be repeated, and they will stay 8 hours again on the site. They will undergo several blood draws, and their medical condition will be monitored. They will also be requested to return to the site on the next day to repeat these assessments.

Interventions:

* Participants will receive SR-878 in a 1-hour long infusion once. The dose will depend on the cohort;
* Participants in the 3rd-6th cohorts will receive LPS injections twice, in a dose of 2 ng/kg body weight.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 18 to 40 years inclusive on the day of informed fonsent form (ICF) signature and with a body weight ≥ 45 kg and body mass index (BMI) ≤ 30 kg/m2;
2. Subjects willing to sign a written informed consent and able to comply with the study protocol for the duration of the study, including the inpatient confinement for about 24 or 32 hours;
3. Has adequate venous access for blood collection;
4. In female subjects of childbearing potential, a negative serum pregnancy test at screening;
5. Females of childbearing potential agreeing to use highly effective methods of contraception for the duration of the study; Males agreeing to use highly effective methods of contraception and not to donate sperm until 90 days after the study drug administration.

Exclusion Criteria:

1. Treatment with an investigational drug within one month or two half-lives prior to screening, whichever is longer;
2. Abnormal findings in medical history and physical examination that the investigator considers to be a clinically relevant abnormality;
3. Clinically significant abnormal screening laboratory tests, including but not limited to:

   * Haemoglobin (HGB) < 120 g/L for males or < 110 g/L for females
   * White Blood Cells (WBC) > 1.5 upper limit of normal (ULN)
   * C-reactive Protein (CRP) > 1.5 ULN
   * Serum Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) or Alkaline Phosphatase (ALP) > 1.5 ULN
   * Estimated Glomerular Filtration Rate (eGFR) < 55 mL/min/1.73 m2
4. Subjects infected with human immunodeficiency virus (HIV), hepatitis B and C viruses (HBV and HCV);
5. Clinically relevant ECG (12 leads) abnormalities;
6. Subjects with acute infectious diseases within 2 weeks prior to screening;
7. History of any autoimmune diseases or any chronic inflammation;
8. Relevant history of other renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine, inflammatory, chronic infectious, or neurological diseases;
9. History of anaphylaxis to drugs or major allergic reactions in general, which in the view of the investigator may compromise the safety of the subjects;
10. Known hypersensitivity to the active substance or to any of the excipients of the investigational medicinal products or auxiliary medicinal products;
11. Drug abuse, alcohol >1 drink/day, defined according to the Food-based Dietary Guidelines in Europe;
12. Females who are pregnant, breastfeeding, or planning to become pregnant during the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Occurrence of treatment-emergent adverse event (TEAE) | Day 1 to Day 85 in Cohorts 1-2 and Day 1 to 86 in Cohorts 3-6
  The number and proportion of subjects with TEAE overall and before the LPS challenge will be calculated by cohort and by arm.

SECONDARY OUTCOMES:
Terminal half-life (T1/2) of SR-878 | Day 1 until Day 85
  Time it takes for the blood plasma concentration of SR-878 to halve its steady-state
Area under the blood concentration-time curve 0-85 days (AUC0-85) | Day 1 until Day 85
  Area under the serum SR-878 concentration versus time curve
AUC0-inf | Day 1 until Day 85
  The area under the plasma SR-878 concentration-time curve extrapolated to infinity
Maximum concentration (Cmax) | Day 1 until Day 85
  Maximum concentration of SR-878 in blood serum
Reference-adjusted area under the effect curve 0-24 hours (AUEC0-24) | 0-24 hours
  The effect of lipopolysaccharide is measured as serum concentrations of tumour necrosis factor-alpha (TNF-alpha).
Maximum effect (Emax) for tumour necrosis factor-alpha (TNF-alpha) after lipopolysaccharide (LPS) challenges | Day 2-3 and Day 85-86
  The maximum effect of lipopolysaccharide is measured as the maximum serum concentrations of tumour necrosis factor-alpha (TNF-alpha).
Safety Measurement Assessment - Adverse Events, including Serious Adverse Events | Day 1 until Day 85 or until day 85 (cohorts 3-6)
  Reports about Adverse Events, including Serious Adverse Events, are collected, standard terms are recorded
Safety Measurement Assessment - Physical Examination | Day 1 until Day 85 or until day 86 (cohorts 3-6)
  Assessment of the head (external), eyes, ears, nose, throat, lungs, cardiovascular system, abdomen, musculoskeletal system, skin, lymph nodes, central nervous system, and, where appropriate, other body systems. Results of assessments are noted as descriptions. There are no units of measurements. There are no individual parameters, the description provides an overall assessment.
Safety Measurement Assessment - Vital signs - Respiratory rate | Screening, Day 1 to day 85 (cohorts 1-2) or to day 86 (cohorts 3-6)
  Breaths per minute
Safety Measurement Assessment - Vital signs - Blood pressure | Screening, Day 1 to day 85 (cohorts 1-2) or to day 86 (cohorts 3-6)
  Pressure or force of blood inside arteries, measured in millimeters of mercury (mmHg).
Safety Measurement Assessment - Vital signs - Heart rate | Screening, Day 1 to day 85 (cohorts 1-2) or to day 86 (cohorts 3-6)
  Frequency of heart beats per minute
Safety Measurement Assessment - Vital signs - Body temperature | Screening, Day 1, 2, 3, 4, 8, 11, and 86 (cohorts 3-6).
  Body temperature is measured °C.
Safety Measurement Assessment - Vital signs - Oxygen saturation | Day 2, day 85
  The unit for oxygen saturation is per cent (%).
Safety Measurement Assessment - Electrocardiogram (ECG) recording | Screening, Day 1, 2, 3, 11, 85, and 86 (cohorts 3-6).
  ECG (12-leads) measuement is used to determine the time intervals for periods of the heartbeat called QRS, QT, and QT interval corrected by Frederic's formula (QTcF)
Safety Measurement Assessment - Urinalysis - Protein concentration | Screening, Day 1, 2, 3, 11, 29, 85 and 86 (cohorts 3-6)
  Protein concentration in urine [mg/dL]
Safety Measurement Assessment - Urinalysis - Blood | Screening, Day 1, 2, 3, 11, 29, 85 and 86 (cohorts 3-6)
  Blood concentration is measured as concentration of hemoglobin
Safety Measurement Assessment - Urinalysis - Glucose concentration | Screening, Day 1, 2, 3, 11, 29, 85 and 86 (cohorts 3-6)
  Glucose concentration in urine as mg/dL
Safety Measurement Assessment - Monitoring of local tolerability | Day 1, 2 and 85
  Assessment of degree of local tolerability in terms of erythema and swelling at the injection site immediately and 1.5 hours after the start of IMP and LPS administration.
Safety Measurement Assessment - Coagulation parameters - INR | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3-6).
  INR = international normalised ratio (which has no dimension)
Safety Measurement Assessment - Coagulation parameters - aPTT | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3-6).
  aPTT = Activated partial thromboplastin time
Safety Measurement Assessment - Coagulation parameters - Fibrinogen | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3-6).
  Concentration of the protein fibrinogen is measured in mg/dL.
Safety Measurement Assessment - Haematology - Haemoglobin | Screening, Day 1, 2, 3, 11, 29, 85, and 86 (cohorts 3 - 6)
  Haemoglobin concentration in blood in g/dL
Safety Measurement Assessment - Haematology - Haematocrit | Screening, Day 1, 2, 3, 11, 29, 85, and 86 (cohorts 3 - 6)
  Percentage of cellular ingredients of blood, measured in per cent (%)
Safety Measurement Assessment - Haematology - Red blood cell count | Screening, Day 1, 2, 3, 11, 29, 85, and 86 (cohorts 3 - 6)
  Number of red blood cells per blood volume
Safety Measurement Assessment - Haematology - White blood cell count | Screening, Day 1, 2, 3, 11, 29, 85, and 86 (cohorts 3 - 6)
  Number of white blood cells per volume blood
Safety Measurement Assessment - Haematology - Platelets | Screening, Day 1, 2, 3, 11, 29, 85, and 86 (cohorts 3 - 6)
  Number of platelets per blood volume
Safety Measurement Assessment - Haematology - Differential blood cell count | Screening, Day 1, 2, 3, 11, 29, 85, and 86 (cohorts 3 - 6)
  Number of neutrophils, eosinophils, basophils, monocytes, lymphocytes per volume blood
Safety Measurement Assessment - Blood chemistry - Potassium | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum concentration of potassium in mmol/L
Safety Measurement Assessment - Blood chemistry - Calcium | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum concentration of calcium in mmol/L
Safety Measurement Assessment - Blood chemistry - Chloride | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum concentration of chloride in mmol/L
Safety Measurement Assessment - Blood chemistry - Sodium | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum sodium concentration in mmol/L
Safety Measurement Assessment - Blood chemistry - Uric acid | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum concentration of uric acid in mmol/L
Safety Measurement Assessment - Blood chemistry - Urea | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum concentration of urea in mmol/L
Safety Measurement Assessment - Blood chemistry - Creatinine | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum concentration of creatinine in μmol/L
Safety Measurement Assessment - Blood chemistry - Total bilirubin | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum concentration of total bilirubin in μmol/L
Safety Measurement Assessment - Blood chemistry - Total protein | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum concentration of total protein in g/L
Safety Measurement Assessment - Blood chemistry - Lactate dehydrogenase | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum concentration of lactate dehydrogenase in U/L
Safety Measurement Assessment - Blood chemistry - Glucose | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum concentration of glucose in mmol/L
Safety Measurement Assessment - Blood chemistry - CRP | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum concentration of CRP = C-reactive Protein in mg/L
Safety Measurement Assessment - Blood chemistry - Alkaline Phosphatase | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum concentration of alkaline phosphatase in U/L
Safety Measurement Assessment - Blood chemistry - Gamma-glutamyl Transferase | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum concentration of gamma-glutamyl transferase in U/L
Safety Measurement Assessment - Blood chemistry - Alanine Aminotransferase | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum concentration of alanine aminotransferase in U/L
Safety Measurement Assessment - Blood chemistry - Aspartate Aminotransferase | Screening, Day 1, 2, 3, 11, 29, 85 and day 86 (cohorts 3 - 6)
  Blood serum concentration of aspartate aminotransferase in U/L

OTHER OUTCOMES:
Levels of tumour necrosis factor-alpha, and their ratios to baseline after SR-878 administration in Cohorts 1-6 | Day 1 until Day 22
  Serum concentration of tumour necrosis factor-alpha on one day of days 1 to 22 divided through serum concentration of tumour necrosis factor-alpha on day 1
Development of anti-drug antibodies | Day 1 - Day 85
  Serum concentration of antibodies against SR-878

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Reeß, Dr., Study Chair — SciRhom GmbH
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to the website of the sponsor of the clinical trial. — https://scirhom.com/